CLINICAL TRIAL: NCT07341243
Title: The Effect of Acute Heat Exposure on Glucose Use During Moderate-intensity Exercise in People With Type 1 Diabetes
Brief Title: Exercising in Hot Conditions: How Does it Effect Blood Glucose in People With T1D
Acronym: T1D-Heat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 25/SPS/065
Record Dates: First submitted 2025-11-25; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: exercise; heat
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temperate (Active Comparator): 40 minutes of moderate intensity continuous exercise at 20°C with 50% relative humidity
  Interventions: Behavioral: Exercise
- Heat (Experimental): 40 minutes of moderate intensity continuous exercise at 40°C with 50% relative humidity
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — exercise in the heat or temperate conditions

SUMMARY:
A randomised, crossover, counterbalanced repeated measures study will be conducted to examine the effect of acute heat exposure on rate of change in blood glucose concentration during 40 minutes of moderate-intensity exercise and for 30 minutes after exercise. Participants will complete two experimental conditions during two separate laboratory visits, with the order of conditions randomised. One condition will be a temperate condition of 20°C with 50% relative humidity (Temperate), the other will be 40°C with 50% relative humidity (Heat). Visits will be identical, including time of day, except for the condition. Visits will be separated by 24h. Testing will take place in the laboratories of the Research Institute for Sport and Exercise Sciences at Liverpool John Moores University.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis more than 1 years ago (to ensure participants are out of the honeymoon period)
* Using insulin therapy with multiple daily injections (MDI), insulin pump (pump), or hybrid closed-loop (HCL)

  o If using a HCL system have experience of using a pre-programmed basal rate in manual mode during exercise
* Aged 18-65 years
* Regularly engaged in endurance exercise (training at least twice per week for ≥30 minutes per session)

Exclusion Criteria:

* Pregnancy
* <6 months postpartum or stopped breastfeeding <1 month before recruitment
* Existing cerebrovascular or cardiovascular disease
* Significant history of hyperglycaemia (HbA1c >85 mmol/mol)
* History of severe hypoglycaemia requiring third party assistance within the last 3 months
* Body weight <36.5kg
* Difficulty swallowing tablets
* Appointment for an MRI test that cannot be rescheduled
* Obstructive gastrointestinal disease
* History of gastrointestinal surgery
* Have an implanted medical device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
blood glucose | Baseline pre exercise to end of exercise (40 minutes)
  change in blood glucose concentration

SECONDARY OUTCOMES:
Core temperature | Baseline pre exercise to end of exercise (40 minutes)
  change in core temperature
Skin temperature | Baseline pre exercise to end of exercise (40 minutes)
  change in skin temperature
Free fatty acids | Baseline pre exercise to end of exercise (40 minutes)
  change free fatty acid concentration
insulin | Baseline pre exercise to end of exercise (40 minutes)
  Change in insulin concentration
glucagon | Baseline pre exercise to end of exercise (40 minutes)
  change in glucagon concentration
epinephrine | Baseline pre exercise to end of exercise (40 minutes)
  change in epinephrine concentration
norepinephrine | Baseline pre exercise to end of exercise (40 minutes)
  change in norepinephrine concentration
cortisol | Baseline pre exercise to end of exercise (40 minutes)
  change in cortisol concentration
Growth hormone | Baseline pre exercise to end of exercise (40 minutes)
  change in Growth hormone concentration
lactate | Baseline pre exercise to end of exercise (40 minutes)
  change in lactate concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
On request to PI